CLINICAL TRIAL: NCT03643185
Title: Cytokine Profile of Allergic Bronchopulmonary Aspergillosis and Its Relevance to Severity and Exacerbation.
Brief Title: Cytokine Profile of Allergic Bronchopulmonary Aspergillosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Director of Respiratory Medicine, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 20180627
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: ABPA
Keywords: cytokine; ABPA; Type 2 immune response; PBMC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage fluid, serum and whole blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main aim of this study is to determine whether the levels of different inflammatory cytokines in the serum and BALF (bronchoalveolar lavage fluid) are relative to the severity and exacerbations of ABPA (allergic bronchopulmonary aspergillosis).

DETAILED DESCRIPTION:
The study would record patients' medical data at baseline and follow them up for different period of time. Updated data would be recorded and blood( or BALF) of the patients would be drawn for tests or stored as whole blood or serum at -80℃ when patients visit the hospital. Then the cytokine (A panel set by the manufacturer) of the serum and BALF would be tested . The secretion ability of peripheral blood mononuclear cells would also be verified. The investigators would then analyze the data and see if any cytokine is relative to the exacerbation or other indicators of the severity of ABPA.

ELIGIBILITY:
For ABPA patients

Inclusion Criteria:

* Patients diagnosed as allergic bronchopulmonary aspergillosis (ABPA). The diagnosis criteria of ABPA is as following: clinical diagnosis of asthma, elevated total IgE levels (> 1,000 IU/mL), presence of specific IgE against A fumigatus detected (> 0.35 kUA/L) or type 1 skin reaction to Aspergillus antigen. Other criteria(at least two of three): Presence of serum IgG antibodies (precipitins) against A. fumigatus; Radiographic pulmonary opacities consistent with ABPA(It might be transient consolidation, nodules, finger-in-glove opacities. Or it could be permanent bronchiectasis and pleuropulmonary fibrosis) Patients who sighed consent forms.

For asthma patients:

Diagnosis according to GINA.

For healthy control:

People with ongoing chronic allergic disease such as allergic rhinitis, asthma and allergic dermatitis are excluded.

Exclusion Criteria:

* Patients who are unwilling to sign the consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ABPA patients who were or would be hospitalized in Shanghai Pulmonary Hospital would be recruited. They would receive standard treatment of ABPA and be asked to visit the clinic again one month later after they start taking glucocorticoids. they are also asked to visit the clinic every three month to monitor the change of serum IgE and their condition. Asthma patients and healthy controls are also enrolled as contrast groups.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2021-05-04 (Estimated); Study Completion 2021-05-04 (Estimated)

PRIMARY OUTCOMES:
Cytokines levels | 1 year
  The levels of different cytokines in the serum or BALF at the enrollment and during follow up. The relation of different cytokines levels and characteristics of ABPA patients would be analyzed.

SECONDARY OUTCOMES:
Exacerbation | 1 year
  The worsening of the symptoms of patients, or the new infiltrate of lung under CT scan that is relevant to ABPA, or the elevated serum IgE level.
High attenuation mucus (HAM) | Once
  It is defined objectively on a CT scan as having an attenuation value > 70 Hounsfield units, visually denser than the paraspinal skeletal muscle
Eosinophilia | 1 year
  Equal to or more than 500/μl
FeNO | 1 year
  The fraction of exhaled nitric oxide
Phenotypes of ABPA | Once
  Patients would be categorized into three phenotypes: ABPA-S (seropositive), ABPA-CB (central bronchiectasis) and ABPA-ORF (other radiologic findings)
Time to exacerbation | 1 year
  The onset date of therapy and the date of the next exacerbation would be recorded to calculate the time to the next exacerbation
Level of different cytokine secreting cells | 1 year
  PBMC would be stained immediately or co-cultured with PMA/ionmycin before staining for flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-fu Xu, MD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China